CLINICAL TRIAL: NCT05506696
Title: A Feasibility Study of Perioperative Vitamin D Supplementation in Patients Undergoing Colorectal Cancer Resection
Brief Title: Vitamin D Supplementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014/0058.1
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Vitamin D Deficiency
Keywords: colorectal; vitamin D
MeSH Terms: conditions — Colorectal Neoplasms; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplementation (Experimental): 3200IU cholecalciferol (Fultium) peri-operatively
  Interventions: Dietary Supplement: Fultium
- Control (No Intervention): No treatment. Control arm.

INTERVENTIONS:
Dietary Supplement: Fultium — 3200IU Fultium
  Arms: Vitamin D supplementation

SUMMARY:
Patients with colorectal cancer will be recruited to undergo vitamin D supplementation in the peri-operative period. Vitamin D levels (25OHD) will be measured to assess response to supplementation.

DETAILED DESCRIPTION:
Patients with a new diagnosis of colorectal cancer will be recruited from colorectal outpatient clinics after confirmation of eligibility. Potential participants will be identified by their healthcare team comprising of clinical nurse specialist or surgeon and co-enrolment with portfolio studies including ALLEGRO and Prepare-ABC will be permitted. Patients undergoing neo-adjuvant therapy, already established on supplementary Vitamin D or with contra-indications to vitamin D supplementation will be excluded. After informed consent participants will undergo blood sampling at baseline (for 25OHD level and DNA) and given 3200IU cholecalciferol (Fultium) per day to take until the time of surgery (median time from pre-operative clinic 4 weeks). Further blood sampling will be performed on the day of surgery, in the early post-operative period (1-2 days, 3-5 days, 6-9 days) and at the first post-operative clinic appointment. Where possible surplus serum from clinically indicated blood tests will be collected to assay 25OHD and reduce need to additional venesection.

ELIGIBILITY:
Inclusion criteria -

* All participants will be aged 16 years or over.
* Participants must be resident in the United Kingdom.
* Undergoing bowel cancer surgery

Exclusion criteria

* Patients who may be at increased risk from Vitamin D supplementation including:
* Kidney disease
* High levels of calcium in the blood
* Atherosclerosis
* Sarcoidosis
* Histoplasmosis
* Over-active parathyroid gland (hyperparathyroidism)
* Lymphoma
* Currently taking thiazide diuretics, digoxin or other cardiac glycosides
* Known allergy to nuts (as peanut oil contained within vitamin D preparations)
* Female subjects of child bearing age who are not taking effective contraception during the period of the trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-09-24 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
25OHD level | Peri-operative, up to 4 weeks post-operative
  25OHD level measured by LC/MS

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Dunlop, Principal Investigator — University of Edinburgh
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No